CLINICAL TRIAL: NCT02364219
Title: Impact of Prewarming on Perioperative Body Core Temperature and the Outcomes of Cytoreductive- and Major Open Abdominal Surgery: A Randomised Trial (PREWARM)
Brief Title: Impact of Prewarming on Perioperative Body Core Temperature and the Outcomes of Cytoreductive- and Major Open Abdominal Surgery: A Randomised Trial
Acronym: PREWARM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Dr. Michael Boschmann, Experimental & Clinical Research Center(ECRC), Charité Berlin-Buch (Unknown)
Responsible Party: Principal Investigator, Michael Sander, Univ.-Prof. M. Sander, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA1/348/14
Record Dates: First submitted 2015-01-20; First posted 2015-02-18 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Hypothermia
Keywords: prewarming; perioperative hypothermia; microdialysis; tissue oxygen saturation; cytoreductive surgery
MeSH Terms: conditions — Hypothermia | interventions — Microdialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard (No Intervention): Study arm in which patients are treated according to standard operating procedures. Acting as "control arm".
- Standard + Microdialysis (Experimental): Study arm in which patients are treated according to standard operating procedures but also receive Microdialysis through a small catheter which is inserted into subcutaneous upper arm fatty tissue.
  Interventions: Device: Microdialysis
- Prewarm (Experimental): Study arm in which patients are treated according to standard operating procedures plus prewarming period of at least 30 minutes during induction of combined general and epidural anesthesia.
  Interventions: Other: Prewarming
- Prewarm + Microdialysis (Experimental): Study arm in which patients are treated according to standard operating procedures plus prewarming period of at least 30 minutes during induction of combined general and epidural anesthesia and Microdialysis through a small catheter which is inserted into subcutaneous upper arm fatty tissue
  Interventions: Other: Prewarming; Device: Microdialysis

INTERVENTIONS:
Other: Prewarming — Patients are treated according to standard operating procedures plus prewarming period of at least 30 minutes during induction of combined general and epidural anesthesia.
  Arms: Prewarm; Prewarm + Microdialysis
Device: Microdialysis — 71 High Cut-Off Brain MD Catheter Membrane cut-off: 100 kDa Membrane length 30 mm Shaft length: 60 mm Dialysis AB, Stockholm, Sweden
  Arms: Prewarm + Microdialysis; Standard + Microdialysis

SUMMARY:
The primary purpose of this study is to determine whether a prewarming period of at least 30 minutes during induction of general and combined epidural anesthesia reduces the core temperature drop normally occuring in patients undergoing cyto-reductive and major abdominal surgery. In addition the effect of prewarming on intra and postoperative body core temperature will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* elective cytoreductive or major abdominal surgery caused by ovarian cancer, primarily or secondary

Exclusion Criteria:

* age < 18
* refusal participate in study
* pregnant or breast-feeding women
* cardiac ejection fraction < 30%
* terminal renal insufficiency requiring dialysis
* severe pulmonary disease (Gina-Classification< 3)
* neurological and/or psychiatric disease
* patient is placed in an institution due to court order
* lack of language skills/understanding
* employee of Charité Berlin
* alcohol addiction
* refusal of epidural anesthesia or failure to insert epidural catheter
* participation in other perioperative, invasive studies which prohibit further study inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
body core temperature drop from induction of anesthesia to start of surgery | approximately 30-40 minutes

SECONDARY OUTCOMES:
body core temperature at the end of surgery | duration of surgery

OTHER OUTCOMES:
prolonged need for ventilatory support | 10 days postoperative
  Goal is to determine whether discrepancies between the different groups regarding prolonged postoperative need for ventilatory support.Defined through length of ventilation after surgery (hours)
Changes in Microcirculation | duration of surgery
  Goal is to determine whether the prewarming and hypothetically improved perioperative warming results in increased microcirculation determined through microdialysis.Measured in lactate/pyruvate (µmol/L) ratio

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sander, Principal Investigator — Department of Anesthesiology and Intensive Care Medicine Campus Charité Mitte / Campus Virchow-Klinikum Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine Campus Charité Mitte / Campus Virchow-Klinikum, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Kaufner L, Niggemann P, Baum T, Casu S, Sehouli J, Bietenbeck A, Boschmann M, Spies CD, Henkelmann A, von Heymann C. Impact of brief prewarming on anesthesia-related core-temperature drop, hemodynamics, microperfusion and postoperative ventilation in cytoreductive surgery of ovarian cancer: a randomized trial. BMC Anesthesiol. 2019 Aug 22;19(1):161. doi: 10.1186/s12871-019-0828-1. PMID 31438849